CLINICAL TRIAL: NCT06900530
Title: Evaluating Sleep Quality With Emerging Technologies
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY20221147
Record Dates: First submitted 2025-02-27; First posted 2025-03-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Snoring; Sleep Disturbances; Hypoxia; Obstructive Sleep Apnea (OSA)
Keywords: Sleep quality; AHI; OSA
MeSH Terms: conditions — Snoring; Parasomnias; Hypoxia; Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Subjects will be given the NOSE Questionnaire, STOP-BANG Questionnaire, SleepCycle app, and Belun Ring. They will be asked to use the equipment for 7 days and report back

SUMMARY:
To investigate the sleep quality of the adult orthodontic patient population at the Case Western Reserve University School of Dental Medicine using the NOSE Questionnaire, STOP-BANG Questionnaire, SleepCycle app, and Belun Ring.

The sample will consist of adult orthodontic patients who came seeking care at the Case Western Reserve University School of Dental Medicine's Orthodontic Department.

Inclusion criteria include adult patients in active treatment in the Case Western Reserve University School of Dental Medicine's Orthodontics Department, age 20 or higher, willingness to give informed consent and participate in the study, possession of a smartphone, and ability to return the Belun Ring and complete the follow-up questionnaire. Exclusion criteria include age less than 20, current or history of taking blood pressure medication, pregnancy, hypovolemia, allergy to thermoplastic elastomers or polycarbonates, anemia, use of mandibular repositioning devices, or active palatal expansion.

There were no existing publications similar to our study found in the current literature. So, the required sample size was estimated by the G Power formula for prevalence studies. The global prevalence of AHI 15 was used to estimate the required sample size for this study. The required sample size for 80% power and .05 precision came to 26 subjects.

DETAILED DESCRIPTION:
Patients will complete four questionnaires (STOP-BANG, NOSE Score, Epworth Sleepiness Scale, and PROMIS Sleep Disturbance Questionnaire), and then wear the Belun Ring for 7 consecutive nights and use the Sleep Cycle App for seven consecutive nights. Patients also will complete a sleep tracking journal. Data points collected by the Belun Ring will include start time, end time, total recording time, oxygen desaturation index, total minutes when spO2 higher than 90%, minimum spO2 percentage, percent of time below 90% O2 saturation, mean spO2, sleep efficiency, bAHI, REM sleep (%), mean pulse rate, and total sleep time. The data collected by the Sleep Cycle will include time in bed, time asleep, minutes snoring, sleep regularity, and sleep quality.

The Sleep Cycle app and the Belun Ring will be used used simultaneously. Ideally, all seven night of the week will have data collected. If the patient skips a night of data collection, they will be encouraged to continue the study regardless.

Microsoft Excel will be used for data analysis. The Jarque Bera test will be used to test for the normality of data distribution. Descriptive statistics will be calculated for each category of data from the questionnaires, Belun Ring, and Sleep Cycle app. Correlation analyses will also be performed between all categories of data. One-way Analysis of Variance (ANOVA) tests will be used to assess whether there are significant differences in the data collected each day of the week for the Belun Ring and Sleep Cycle app, at the p=0.05 level of statistical significance. One-way T-tests will be used to compare data between subjects with bAHI less than 10 and bAHI higher than 10.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 75 years of age
* Current orthodontic patient at Case Western Reserve University
* Possession of a smartphone
* Ability to return Belun ring

Exclusion Criteria:

* Less than 20 or older than 75 years of age.
* Current or history of taking blood pressure medication, pregnancy, hypovolemia, allergy to thermoplastic elastomers or polycarbonates, anemia, use of mandibular repositioning devices, or active palatal expansion.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult orthodontic patients
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Nasal Obstruction Assessment (NOSE) Questionnaire Score | baseline
  The NOSE questionnaire is a validated tool that assesses nasal blockage. It provides an objective score that ranges from 0 to 100 with lower scores indicating less nasal blockage and higher scores indicating worse nasal blockage.
Adult Obstructive Sleep Apnea (STOPBAng) Questionnaire | baseline
  The STOPBang questionnaire is a validated tool that assesses the risk of obstructive sleep apnea (OSA). It provides an objective score that ranges from 0 to 8 with lower scores indicating lower risk of sleep apnea and higher scores indication higher risk of sleep apnea.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Questionnaire | baseline
  The PROMIS Sleep Disturbance Questionnaire assesses the quality of sleep objectively that ranges from 8 to 40 with lower scores indicating less sleep disturbance and higher scores indicating more severe sleep disturbances.
Epworth Sleepiness Scale (ESS) Questionnaire | baseline
  The Epworth Sleepiness Scale Questionnaire is a validated tool to assess daily sleepiness. It provides an objective score that can range from 0 to 24 with lower scores indicating less daytime sleepiness and higher scores indicating more severe daytime sleepiness.
Belun Ring REM sleep percentage. | The subject is asked to use it for 7 days, and the average and standard deviation of those 7 days is the outcome that will be used.
  The Belun ring measures the the mean REM sleep percentage.
Belun Ring Oxygen Saturation | The subject is asked to use it for 7 days, and the average and standard deviation of those 7 days is the outcome that will be used.
  The Belun ring measures the mean oxygen saturation as the average percentage of oxygen saturation in the blood.
Belun Ring apnea/hypopnea index | The subject is asked to use it for 7 days, and the average and standard deviation of those 7 days is the outcome that will be used.
  The Belun ring measures the apnea/hypopnea index. The outcome is the number of apneic events per hour of sleep.
SleepCycle App | The subject is asked to use it for 7 days, and the average and standard deviation of those 7 days is the outcome that will be used.
  The Sleep Cycle app is a smartphone app that measures time in bed, time asleep, and the presence of snoring.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Palomo, DDS, MSD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University Dental Clinic - Orthodontics, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data without PHI will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study completion
Access Criteria: Upon request

REFERENCES:
- [Background] Schutte-Rodin S, Deak MC, Khosla S, Goldstein CA, Yurcheshen M, Chiang A, Gault D, Kern J, O'Hearn D, Ryals S, Verma N, Kirsch DB, Baron K, Holfinger S, Miller J, Patel R, Bhargava S, Ramar K. Evaluating consumer and clinical sleep technologies: an American Academy of Sleep Medicine update. J Clin Sleep Med. 2021 Nov 1;17(11):2275-2282. doi: 10.5664/jcsm.9580. No abstract available. PMID 34314344
- [Background] Yeh E, Wong E, Tsai CW, Gu W, Chen PL, Leung L, Wu IC, Strohl KP, Folz RJ, Yar W, Chiang AA. Detection of obstructive sleep apnea using Belun Sleep Platform wearable with neural network-based algorithm and its combined use with STOP-Bang questionnaire. PLoS One. 2021 Oct 11;16(10):e0258040. doi: 10.1371/journal.pone.0258040. eCollection 2021. PMID 34634070
- [Background] Gu W, Leung L, Kwok KC, Wu IC, Folz RJ, Chiang AA. Belun Ring Platform: a novel home sleep apnea testing system for assessment of obstructive sleep apnea. J Clin Sleep Med. 2020 Sep 15;16(9):1611-1617. doi: 10.5664/jcsm.8592. PMID 32464087
- [Background] Nagappa M, Liao P, Wong J, Auckley D, Ramachandran SK, Memtsoudis S, Mokhlesi B, Chung F. Validation of the STOP-Bang Questionnaire as a Screening Tool for Obstructive Sleep Apnea among Different Populations: A Systematic Review and Meta-Analysis. PLoS One. 2015 Dec 14;10(12):e0143697. doi: 10.1371/journal.pone.0143697. eCollection 2015. PMID 26658438
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Klaus K, Stummer AL, Ruf S. Accuracy of a Smartphone Application Measuring Snoring in Adults-How Smart Is It Actually? Int J Environ Res Public Health. 2021 Jul 8;18(14):7326. doi: 10.3390/ijerph18147326. PMID 34299777
- [Background] Figueras-Alvarez O, Canto-Naves O, Cabratosa-Termes J, Roig-Cayon M, Felipe-Spada N, Tomas-Aliberas J. Snoring intensity assessment with three different smartphones using the SnoreLab application in one participant. J Clin Sleep Med. 2020 Nov 15;16(11):1971-1974. doi: 10.5664/jcsm.8676. PMID 32638700

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT06900530/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT06900530/ICF_001.pdf